CLINICAL TRIAL: NCT06271603
Title: Evaluation of the Efficiency and Economic Impact of LC-OCT (Line-field Confocal Optical Coherence Tomography) for the Diagnosis and Management of Basal Cell Carcinomas (ECOBASO)
Brief Title: Evaluation of the Efficiency and Economic Impact of LC-OCT (Line-field Confocal Optical Coherence Tomography) for the Diagnosis and Management of Basal Cell Carcinomas
Acronym: ECOBASO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Damae Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23.02645.000357-MS01; CPP Ile de France III (Other: 23.02645.000357-MS01)
Record Dates: First submitted 2024-02-08; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Basal Cell Carcinoma of the Skin
Keywords: basal cell carcinoma diagnosis; LC-OCT
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm: Management performed with an initial diagnosis based on the LC-OCT device (Experimental): The interventional procedure involves the management of BCC with an initial diagnosis based on the deepLive™ device. The imaging is performed by placing the probe tip in contact with the patient's skin after applying an immersion oil (paraffin) to the imaging area. The examination lasts only a few minutes and is painless. An integrated dermoscopic targeting system allows the operator to ensure proper positioning of the probe on the lesion and to ensure that the entire lesion has been captured for an accurate diagnosis. The images are displayed in real-time during the examination and directly evaluated by the investigator, who has the option to save images/videos at their discretion. A final evaluation with the deepLive™ device will also be performed during the 1-year follow-up, and intermediate evaluations may also be performed with the deepLive™ device depending on the initial management of BCC.
  Interventions: Diagnostic Test: diagnosis based on deepLive™ LC-OCT device
- Control Arm: Standard management with an initial diagnosis based on skin biopsy (Active Comparator): The control procedure corresponds to standard management of BCC with an initial diagnosis based on skin biopsy (standard management arm). The biopsy will be performed according to the standard practice of each center, using a 2 to 6 mm punch or shave biopsy, with prior injection of a local anesthetic. A final evaluation with the deepLive™ device will also be performed during the 1-year follow-up.
  Interventions: Diagnostic Test: diagnosis based on skin biopsy

INTERVENTIONS:
Diagnostic Test: diagnosis based on deepLive™ LC-OCT device — Management of BCC with an initial diagnosis based on the deepLive™ device using LC-OCT technology.
  Other Names: LC-OCT arm
  Arms: Intervention Arm: Management performed with an initial diagnosis based on the LC-OCT device
Diagnostic Test: diagnosis based on skin biopsy — Control Arm: Standard management with an initial diagnosis based on skin biopsy
  Other Names: biopsy arm
  Arms: Control Arm: Standard management with an initial diagnosis based on skin biopsy

SUMMARY:
This is a comparative, randomized, prospective, multicenter clinical investigation aimed at evaluating the efficiency and economic impact of LC-OCT (Line-field Confocal Optical Coherence Tomography) for the diagnosis and management of basal cell carcinomas.

DETAILED DESCRIPTION:
Basal cell carcinoma (BCC) is the most common type of skin cancer. The diagnosis and subtyping of suspicious lesions can be challenging for certain "equivocal" lesions where clinical and dermoscopic criteria do not allow for a definite diagnosis or subtyping, which determines the treatment. The most commonly used technique for the diagnosis and selection of appropriate treatment for BCC is skin biopsy. Microscopic imaging techniques allow for "optical" biopsies, which appear as an attractive alternative to traditional biopsies.

The deepLive™ device integrates LC-OCT (Line-field Confocal Optical Coherence Tomography), which is a novel microscopic imaging technology with unmatched imaging performance to date, including cellular isotropic resolution (1 μm), a penetration depth of 500 μm, and the ability to obtain real-time cross-sectional and 3D images in the same orientation as histology. Numerous multicenter studies have confirmed the high performance of this technique for the diagnosis and subtyping of BCC. However, its usefulness in the diagnostic and treatment management of BCC has not been investigated prospectively. This clinical investigation is based on the hypothesis that the use of the deepLive™ device will enable diagnostic and therapeutic management by reducing the number of consultations/procedures without compromising patient outcomes compared to a traditional management approach with biopsy(ies). This strategy could optimize the entire care pathway by reducing invasive diagnostic or therapeutic procedures and freeing up dermatological resources for other procedures. This optimization of the care pathway is expected to result in a favorable economic impact on the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

Patient with one or more clinically suspicious lesions of BCC for which:

1. The diagnosis is uncertain following clinical and dermoscopic examination, and diagnostic biopsy is necessary according to the latest European guidelines from EADO.
2. And/or for which the knowledge of the histological subtype determines the subsequent management.
3. And/or for which diagnostic biopsy is necessary in the standard practice to confirm the clinical diagnosis (peri-orificial facial lesions, any lesion that may require complex surgical reconstruction).

Exclusion Criteria:

* The lesion is suspected to be a recurrent BCC.
* The suspicious lesion has been previously treated by other surgical or non-surgical methods (cryotherapy, topical treatment, PDT, etc.).
* Lesions within 3 cm of the eye.
* Presence of cutaneous comorbidities that could interfere with a proper evaluation of the studied lesion according to the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 704 (Estimated)
Dates: Start 2024-02-26 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to demonstrate, at 1 year, the clinical non-inferiority and organizational and economic superiority of the management of primary BCC through diagnosis with LC-OCT compared to traditional management. | from enrollment to the 1 year follow up
  The primary objective is defined by a family of primary criteria that will be tested sequentially in a hierarchical manner. The clinical non-inferiority will be assessed by the proportion of success which is defined as the absence of residual or recurrent cancerous or precancerous lesions after 1 year of primary BCC through diagnosis with LC-OCT, as compared to traditional management.
The primary objective is to demonstrate, at 1 year, the clinical non-inferiority and organizational and economic superiority of the management of primary BCC through diagnosis with LC-OCT compared to traditional management. | from enrollment to the 1 year follow up
  The primary objective is defined by a family of primary criteria that will be tested sequentially in a hierarchical manner. Organizational effectiveness will be evaluated by measuring the total time spent by dermatologists and pathologists (in hours) for managing primary BCC through diagnosis with LC-OCT, as compared to traditional management.
The primary objective is to demonstrate, at 1 year, the clinical non-inferiority and organizational and economic superiority of the management of primary BCC through diagnosis with LC-OCT compared to traditional management. | from enrollment to the 1 year follow up
  The primary objective is defined by a family of primary criteria that will be tested sequentially in a hierarchical manner. Economic superiority will be assessed by comparing the total cost of management (€) of primary BCC through diagnosis with LC-OCT to traditional management.

SECONDARY OUTCOMES:
Compare, after the diagnosis announcement and at 1 year, the quality of life of patients in the LC-OCT arm versus the standard management arm. | from enrollment to the 1 year follow up
  Quality of life will be assessed using the EQ-5D-5L questionnaire
Compare, after the diagnosis announcement and at 1 year, the anxiety levels of patients in the LC-OCT arm versus the standard management arm. | from enrollment to the 1 year follow up
  Anxiety will be assessed using a visual analog scale (score 0 - 10)
Compare patient satisfaction with their management at 1 year in the LC-OCT arm versus the standard management arm. | from enrollment to the 1 year follow up
  Patient satisfaction will be evaluated using a Likert scale focused on the overall management of the cutaneous lesion.
Evaluate the performance of LC-OCT for the diagnosis and subtyping of BCC for all patients operated on or biopsied in the LC-OCT arm. | from enrollment to the 1 year follow up
  Performance will be evaluated based on the sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), positive likelihood ratio (PLR), negative likelihood ratio (NLR), and accuracy of LC-OCT for the diagnosis and subtyping of BCC in all patients operated on or biopsied in the LC-OCT arm, using histological diagnosis as the gold standard.
Compare dermatologists' satisfaction with patient management in the LC-OCT arm versus the standard management arm | from enrollment to the 1 year follow up
  Physician satisfaction will be evaluated using a Likert scale focused on the overall management of the cutaneous lesion.
Estimate the actual cost of conducting the diagnosis with LC-OCT technology. | from enrollment to the 1 year follow up
  Actual cost (€) of conducting the diagnosis with deepLive™ measured using micro-costing methodology
Compare healthcare consumption between the two groups at 1 year. | from enrollment to the 1 year follow up
  Typology of healthcare consumption at 1 year in each group to identify differences between the two groups in terms of: consultations, treatments, hospitalizations, medical procedures, laboratory tests, imaging, etc.
Conduct a cost-consequence analysis of patient management with LC-OCT technology versus standard management. | from enrollment to the 1 year follow up
  The descriptive cost-consequence analysis will analyze the difference in patient management costs at 1 year in relation to the impacts of deepLive™ on other clinical and organizational criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Ambroise Paré, Boulogne-Billancourt, France